CLINICAL TRIAL: NCT05163613
Title: Use of Low-frequency Magnetic Fields in the Hybrid Treatment of COVID-19 Patients: Preliminary Reports.
Brief Title: Use of Low-frequency Magnetic Fields in the Hybrid Treatment of COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RNN/339/20/KE; RNN/339/20/KE (Other: Bioethics Committee, Medical University)
Record Dates: First submitted 2021-12-17; First posted 2021-12-20 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; COVID-19 Respiratory Infection; COVID-19 Pneumonia
Keywords: COVID-19; magnetostimulation; interleukin; treatment
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with COVID - 19, who we were treated with magnetic stimulation. (Experimental): The study group included patients hospitalized due to PCR-confirmed SARS-Cov-2 infection, who were treated with magnetic stimulation in addition to a standard therapy.
  Standard therapy used in all patients consisted of the use of pharmacological agents necessary to treat the viral infection (antiviral drugs, antibiotics, dexamethasone) and the inclusion of proper care, education, occupational therapy, self-service learning, breathing exercises and motor mobilization.
  Interventions: Other: magnetostimulation; Other: standard therapy
- Patients with COVID - 19, who we were treated without magnetic stimulation. (Experimental): The control group included patients receiving a comprehensive treatment without magnetic stimulation. The patients were in a moderately severe condition.
  Interventions: Other: standard therapy

INTERVENTIONS:
Other: magnetostimulation — Treatment parameters: 12 minutes M2P2 program, with increasing intensity from 1 to 8. The authors applied magnetic field with a frequency of 180 - 190 Hz, pulse packet frequencies between 12.5 and 29 Hz, packet groups 2.8 - 7.6 Hz, series 0.08 - 0.3 Hz, with magnetic induction B= 3.2 µT (on average) and B = 40 µT at a pulse peak.
  Other Names: low frequency magnetic field; magnetostimultaion
  Arms: Patients with COVID - 19, who we were treated with magnetic stimulation.
Other: standard therapy — Standard therapy used in all patients consisted of the use of pharmacological agents necessary to treat the viral infection (antiviral drugs, antibiotics, dexamethasone) and the inclusion of proper care, education, occupational therapy, self-service learning, breathing exercises and motor mobilization.

SUMMARY:
The purpose of this study was to evaluate the efficacy of low-frequency magnetic field in the hybrid treatment of COVID-19 patients, i.e., including magnetostimulation in the standard treatment. The authors evaluated among other things, the immunocorrective therapeutic effect of magnetostimulation, improving the defensive functions of the immune system and thus supporting the immune function by, among other things, suppressing the "cytokine storm".

After application of low-frequency magnetic field in the hybrid treatment of COVID-19 patients, the authors expected: a decrease in the level of proinflammatory factors (IL - 6), restoration of homeostasis in the body with regards to the range of parameters evaluated in laboratory tests (WBC, MONO, PLT, CRP, d-dimers) and normalization of the following parameters: arterial blood pressure, the number of breaths/min, saturation, temperature.

DETAILED DESCRIPTION:
Study aim:

The purpose of this study was to evaluate the efficacy of low-frequency magnetic field in the hybrid treatment of COVID-19 patients, i.e., including magnetostimulation in the standard treatment.

Material and methods:

The study was conducted on patients aged 39 to 80 years, of both sexes affected by COVID-19. The study subjects were recruited at the Covid Unit of the Military Medical Academy University Teaching Hospital - Central Veterans' Hospital in Lodz. The study group (13 patients) included patients hospitalized due to PCR (polymerase chain reaction)-confirmed SARS (severe acute respiratory syndrome) -Cov-2 infection, who were treated with magnetostimulation in addition to a standard therapy. The control group (10 patients) included patients receiving a comprehensive treatment without magnetostimulation. The patients hospitalized due to PCR-confirmed SARS - Cov - 2 infection were qualified for the study. Patients with absolute contraindications to magnetic field application and patients with limited verbal - logical contact were excluded from the study.

In the study groups, the patients were subjected to magnetic field - magnetostimulation with the use of apparatus Viofor JPS System (mata). 14 treatments were performed, 7 times a week. Treatment parameters: 12 minutes M2P2 program, with increasing intensity from 1 to 8. The authors applied magnetic field with a frequency of 180 - 190 Hz, pulse packet frequencies between 12.5 and 29 Hz, packet groups 2.8 - 7.6 Hz, series 0.08 - 0.3 Hz, with magnetic induction B= 3.2 µT (on average) and B = 40 µT at a pulse peak.

In laboratory tests, the following levels were assessed in the patients: interleukin 6 (IL -6), leukocytes (WBC), monocytes (MONO), platelets (PLT), CRP and d-dimers. The patients' blood was taken twice: on admission to the department and after a series of treatments with magnetostimulation. Approximately 6 ml of blood was collected at one time (3 tubes).

Medical records of the patients and scientific reports collected from the University Library and medical databases, e.g. PubMed, were analyzed and discussed.

ELIGIBILITY:
Inclusion Criteria:

- patients hospitalized due to PCR-confirmed SARS - Cov - 2 infection

Exclusion Criteria:

* patients with absolute contraindications to magnetic field application
* patients with limited verbal - logical contact were excluded from the study

Ages: 39 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
the level of proinflammatory factors (IL - 6) | 14 days
  decrease in the level of proinflammatory factors (IL - 6)
the level of leukocytes (WBC) | 14 days
  restoration of homeostasis in the body with regards to the range of WBC
the level of monocytes (MONO) | 14 days
  restoration of homeostasis in the body with regards to the range of MONO
the level of platelets (PLT), | 14 days
  restoration of homeostasis in the body with regards to the range of PLT
the level of CRP (c reactive protein) | 14 days
  restoration of homeostasis in the body with regards to the range of CRP
the level of d-dimers. | 14 days
  restoration of homeostasis in the body with regards to the range of d-dimers
arterial blood pressure, | 14 days
  normalization of the arterial blood pressure,
the number of breaths/min | 14 days
  normalization of the number of breaths/min
saturation | 14 days
  normalization of saturation
temperature | 14 days
  normalization of temperature

CONTACTS AND LOCATIONS:
Overall Officials: Marta Woldańska-Okońska, profesor, Study Director — Department of Rehabilitation and Physical Medicine, Medical University of Lodz; Agnieszka Jankowska, doctor, Principal Investigator — Department of Rehabilitation and Physical Medicine, Medical University of Lodz; Robert Irzmański, profesor, Principal Investigator — Department of Internal Medicine and Cardiac Rehabilitation; Katarzyna Glibov, doctor, Principal Investigator — Department of Internal Medicine and Cardiac Rehabilitation
Locations (1):
- Department of Rehabilitation and Physical Medicine, Medical University of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No